CLINICAL TRIAL: NCT00392197
Title: Post Marketing Clinical Study of Aripiprazole in Patients With Schizophrenia - Effects on Glucose Metabolism-
Brief Title: Study of Aripiprazole in Patients With Schizophrenia- Effects on Glucose Metabolism-
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-05-002-C; JapicCTI-060325
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: OPC-14597; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 1 or 2 times a day, p.o., 6 - 24mg a day
  Other Names: Abilify

SUMMARY:
The objective of this study is to examine the effects of aripiprazole on glucose metabolism in schizophrenic patients without hyperglycemia and diabetes mellitus or any history thereof.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients who are 16 years or older when written informed consent was obtained.
2. Patients who give personal written informed consent to participate in this study.
3. Patients who meet any of the following criteria for antipsychotic-naive or currently antipsychotic-free patients or patients who have been treated with antipsychotics indicated for schizophrenia from the onset of schizophrenia until the time of giving informed consent.

   Antipsychotic-naive or currently antipsychotic-free patients
   * Patients who do not take any antipsychotics
   * Patients who have taken antipsychotics for less than 2 years and discontinued them for 12 weeks prior to giving informed consent

   Patients recently treated with antipsychotics
   * Patients who have taken antipsychotics for more than 2 years and are taking antipsychotics at the time of giving informed consent
4. Patients who meet all of the following conditions

   * Patients who do not have any obvious complication of diabetes mellitus
   * Patients who do not have any obvious medial history with antidiabetic agents
   * Patients with no obvious history of diabetes mellitus recorded in the current charts of the study site at the time of giving informed consent
   * Patients who have not shown any values for the following parameters that deviate from the standard laboratory values in the current charts of the study site at the time of giving informed consent
   * Patients whose laboratory values meet all of the following criteria in the clinical laboratory tests conducted after patients give informed consent, just before commencement of study drug administration.

     * Fasting blood glucose level (FBS) <110mg/dL (If FBS is not available, non-fasting blood glucose level*1 <140mg/dL)

       *1 : For cases in which blood sugar measurements include values that cannot be judged as having been obtained in the fasted state.
     * HbA1c <5.8% Fasting blood glucose is defined as glucose concentrations in plasma samples taken between 5 a.m. and 12 noon after at least eight hours of fasting (including abstinence from snacks and calorie-containing juice, coffee, etc. ). All other blood glucose measurements of are counted random glucose.
5. Patients who have no obvious family history (in parents or siblings) of diabetes mellitus at the time of commencement of study drug administration
6. Patients whose body mass index (BMI) is less than 25 kg/m2 in the current charts of the study site at the time of giving informed consent Body Mass Index (BMI) = Body weight in kg /(height in m)2

Exclusion Criteria:

1. Patients who have been given aripiprazole after market launching
2. Patients who clearly experienced symptoms of polydipsia, including so-called PET-bottle syndrome (hyperglycemia caused when the supply of insulin, which promotes glucose metabolism, becomes insufficient due to continuous soft drink consumption) and water intoxication, within one year prior to giving informed consent
3. Patients taking drugs that affect glucose metabolism
4. Patients who take quetiapine fumarate (Seroquel) or olanzapine (Zyprexia) within a period from 12 weeks prior to commencement of study drug administration to immediately before commencement of study drug administration
5. Patients with the following complications Abnormal adrenal function, abnormal pituitary function, abnormal thyroid function, chronic pancreatitis, chronic hepatitis, alcoholic hepatopathy, non-alcoholic fatty liver, and liver cirrhosis
6. Female patients who are known to have given birth to a macrosomatic infant exceeding 4000 g in weight
7. Patients given antipsychotics at doses equivalent to 20 mg/day or more of haloperidol (or, in the case of multi-drug therapy, a combined equivalence of 20 mg/day or more of haloperidol) within a period from 12 weeks prior to commencement of study drug administration to immediately before commencement of study drug administration
8. Patients in a major state of excitation or stupor immediately before commencement of study drug administration
9. Patients who are forcibly hospitalized
10. Patients given any investigational new drugs within 12 weeks prior to commencement of study drug administration
11. Patients diagnosed as having a complication of serious hepatic, renal, cardiac, or haematopoietic disorder within 4 weeks prior to commencement of study drug administration, according to the criteria specified below.

    Hepatic disorder: Total bilirubin ≥ 3.0 mg/dL, AST (GOT) and ALT (GPT) ≥2.5 times the upper limits of normal levels at the study site.

    Renal disorder: Creatinine ≥ 2 mg/dL Heart: Congestive heart failure arrhythmias, and ischemic heart disease being treated by drug therapy Haematopoietic disorder, etc.: RBC < 3,000,000, Hb <10.0 g/dL, WBC < 3,000, platelet counts < 7,500
12. Pregnant or lactating women, women shown to be possibly pregnant by the pregnancy examination conducted immediately before commencement of study drug administration, and women who are hoping to become pregnant within one year after providing informed consent to participate in the study
13. Patients who meet any of the criteria for contraindication listed on the package insert of aripiprazole
14. Patients with a complication or history of neuroleptic malignant syndrome or a related condition
15. Patients suffering physical exhaustion associated with dehydration or malnutrition, etc.
16. Patients with a complication or history of paralytic ileus
17. Patients with a history of alcohol dependence or drug abuse
18. Patients with a history of suicide attempt, or patients who have a high possibility of committing self-injury or attempting suicide
19. Patients with a complication or history of convulsion disorders, such as epilepsy, or structural brain disorders
20. Patients considered in the judgment of the principal investigator or the attending investigator to be inappropriate for inclusion in the study for any other reason

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Division of New Product Evaluation and Development
Locations (5):
- Japan (5):
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Touhoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Antipsychotic-naïve Patients: Patients who have never taken antipsychotic drugs or patients who have taken antipsychotic drugs for less than 2 years and have not taken them within a period from at least 12 weeks prior to giving informed consent to immediately before commencement of study drug administration
- Patients Previously Treated With Antipsychotic Drugs: Patients who have taken antipsychotic drugs for 2 years or more and are taking antipsychotic drugs at the time of giving informed consent
Period: Overall Study
Arm/Group | Antipsychotic-naïve Patients | Patients Previously Treated With Antipsychotic Drugs
Started | 48 | 63
Completed | 27 | 33
Not Completed | 21 | 30
Not completed — Adverse Event | 4 | 12
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Protocol Violation | 7 | 5
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Population: The glucose metabolism analysis set.
  The numbers of excluded subjects from the data of partcipant flow were:
  * violation of inclusion/exclusion criteria: naïve arm- 4, prior treated arm- 1
  * no data of blood glucose level after treatment: naïve arm- 3, prior treated arm- 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Antipsychotic-naïve Patients | Patients Previously Treated With Antipsychotic Drugs | Total
Number analyzed (Participants) | 43 | 58 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (13.6) | 39.9 (14.0) | 35.7 (14.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 0 | 6
  Between 18 and 65 years | 36 | 54 | 90
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 21 | 29 | 50
Region of Enrollment [Number; unit: participants]
  Japan | 43 | 58 | 101

OUTCOME MEASURES:

1. Primary Outcome: Fasting Blood Glucose (FBS) Level (if Fasting Blood Glucose Level Was Not Available, Non-fasting Blood Glucose (Non-FBS) Level)
Description: The number of subjects whose FBS level reached or exceeded 126 mg/dL (200 mg/dL, non-FBS level) at least once during the test product administration period as well as the incidence were determined. Also, for 110 mg/dL and above (140 mg/dL, non-FBS level), the number of subjects were determined in the same way.
Time Frame: Prior to the start of administration (Baseline) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 52, or discontinuation
Population: Subjects who were treated with at least 1 tablet of the test product, and whose blood glucose level was measured at least once after test product administration were included in the glucose metabolism analysis set. However, subjects who violated inclusion criteria and exclusion criteria were excluded.
Measure: Number; unit: participants
Arm/Group | Antipsychotic-naïve Patients | Patients Previously Treated With Antipsychotic Drugs
Number analyzed (Participants) | 43 | 58
participants
  FBS: 126 mg/dL or above | 0 | 0
  FBS: 110 mg/dL or above | 1 | 4
  non-FBS: 200 mg/dL or above | 0 | 0
  non-FBS: 140 mg/dL or above | 0 | 1

2. Secondary Outcome: HbA1c
Description: The number of subjects with an HbA1c value of 6.5% or higher were calculated. In addition, for 5.8% and above, the number of subjects were also calculated, in the same way
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 52, or discontinuation
Measure: Number; unit: participants
Arm/Group | Antipsychotic-naïve Patients | Patients Previously Treated With Antipsychotic Drugs
Number analyzed (Participants) | 43 | 58
participants
  6.5 % or more increase in HbA1c | 0 | 0
  5.8 % or more increase in HbA1c | 0 | 0

ADVERSE EVENTS:
Time Frame: 54 weeks
Arm/Group | Antipsychotic-naïve Patients | Patients Previously Treated With Antipsychotic Drugs
Serious Adverse Events (participants affected / at risk) | 4/48 | 6/63
Other Adverse Events (participants affected / at risk) | 45/48 | 55/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antipsychotic-naïve Patients (N=48) | Patients Previously Treated With Antipsychotic Drugs (N=63)
Asthenia (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Psychiatric Symptom (Nervous system disorders) | 1 (1) | 4 (4)
Restlessness (Nervous system disorders) | 0 (0) | 1 (2)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antipsychotic-naïve Patients (N=48) | Patients Previously Treated With Antipsychotic Drugs (N=63)
Abdominal Discomfort (Gastrointestinal disorders) | 4 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (11) | 5 (7)
Dental Caries (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 13 (17) | 18 (21)
Alanine Aminotransferase Increased (Investigations) | 4 (4) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 2 (2) | 9 (10)
Blood Prolactin Decreased (Investigations) | 19 (19) | 27 (27)
White Blood Cell Count Decreased (Investigations) | 3 (3) | 2 (2)
Weight Decreased (Investigations) | 0 (0) | 6 (6)
Weight Increased (Investigations) | 11 (11) | 7 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Akathisia (Nervous system disorders) | 16 (17) | 4 (5)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dystonia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Parkinsonism (Nervous system disorders) | 5 (5) | 1 (1)
Somnolence (Nervous system disorders) | 9 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 13 (14)
Psychiatric Symptom (Psychiatric disorders) | 1 (1) | 4 (4)
Restlessness (Psychiatric disorders) | 3 (3) | 1 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 1 (2)
Orthostatic Hypotension (Vascular disorders) | 4 (5) | 0 (0)
Malaise (General disorders) | 3 (3) | 3 (3)
Thirst (General disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No